CLINICAL TRIAL: NCT06788470
Title: Safety and Efficacy of Umbilical Cord-derived Mesenchymal Stem Cell Transplantation in the Treatment of Bronchopulmonary Dysplasia in Premature Infants
Brief Title: Safety and Efficacy of Umbilical Cord-derived Mesenchymal Stem Cell(MSC) Transplantation in the Treatment of Bronchopulmonary Dysplasia(BPD) in Premature Infants
Acronym: MSC，BPD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Shu Qiang, Professor of Pediatrics, Chief surgeon, Principal Investigator, Hospital secretary of Party Committee, Children's Hospital, Zhejiang University School of Medicine, The Children's Hospital of Zhejiang University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-SC-001
Record Dates: First submitted 2025-01-06; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: BPD - Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary dysplasia (BPD); Mesenchymal stem cells (MSCs); Premature infants
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Intervention Model Description: Intratracheal administration of umbilical cord-derived mesenchymal stem cells (MSCs) in premature infants with bronchopulmonary dysplasia (BPD).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MSC transplantation (Experimental): MSCs (1×10^7/kg) are administered intratracheally to participators.
  Interventions: Drug: MSC

INTERVENTIONS:
Drug: MSC — Intratracheal administration of umbilical cord-derived mesenchymal stem cells (MSCs).

SUMMARY:
Bronchopulmonary dysplasia (BPD) is a chronic lung disease, which is a major complication of very low and ultra-low preterm infants. Moderate and severe BPD survivors are prone to adverse outcomes such as impaired lung function, childhood exercise intolerance, and neurodevelopmental retardation in the long term, which seriously affects their quality of life and brings a heavy burden to society and families. However, the pathogenesis of BPD is complex, including pulmonary vascular dysplasia, lung inflammation, and impaired alveolar development. There is currently no specific clinical drug to cure BPD. Mesenchymal stem cells (MSCs) are a kind of multipotent stem cells that exist in almost all organs and tissues of individuals. MSCs have the properties including self-renewal, multi-directional differentiation, and immunosuppressive and anti-inflammatory abilities. Preclinical studies have shown that MSCs can alleviate BPD by improving alveolar and pulmonary vascular development, and reducing pulmonary fibrosis. Several phase I clinical studies have demonstrated that intratracheal transplantation of human umbilical cord blood-derived mesenchymal stem cells for children with BPD is safe and feasible.

This study aims to further evaluate the safety and efficacy of umbilical cord-derived mesenchymal stem cell transplantation in the treatment of severe BPD in premature infants, in the hope of increasing the survival rate and improving the prognosis of severe BPD.

ELIGIBILITY:
Inclusion Criteria:

1. 23-29 weeks of gestation, birth weight 500-1500g;
2. For patients with no improvement or aggravation of lung condition after DART hormone therapy, and positive pressure ventilation by tracheal intubation is still required at a correct gestational age of 36 weeks.
3. Children with severe BPD after early use of PS
4. Parents agree to participate in clinical trials.

Exclusion Criteria:

1. Premature infants not suitable for the given gestational age;
2. Other congenital structural malformations of trachea, bronchus and lungs;
3. Complicated with severe congenital heart disease;
4. Complicated with Periventricular Leukomalacia (PVL);
5. Complicated with intraventricular hemorrhage (IVH) above level 3;
6. Septic shock or positive blood culture;
7. Acute pulmonary hemorrhage;
8. Intracranial and extracranial diseases affecting respiratory rate and rhythm.

Min Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2027-08-09 (Estimated); Study Completion 2027-08-09 (Estimated)

PRIMARY OUTCOMES:
Extubating time after MSC transplantation | until 24 months of corrected age
  Record how long it takes for the participants' tracheal tubes to be removed after MSC transplantation.
The number of times and total duration of re-intubation after extubating | until 24 months of corrected age
  If the participants' tracheal tubes are removed after MSC transplantation, record the number of times and total duration of tracheal re-intubation until discharge and 24 months of corrected age.
Mortality of BPD | until 24 months of corrected age
  Record the number of participants who died from BPD.

SECONDARY OUTCOMES:
Further assess the severity of BPD by detecting the levels of pro-inflammatory cytokine in alveolar lavage fluid, pulmonary function index and chest radiography. | until 24 months of corrected age
  The levels of pro-inflammatory cytokine (IL-6, IL-8, TNF-α, IL-1β, IL-10, MMP-9, TGF-β) in alveolar lavage fluid are examined via ELISA kits before and at 7 days after MSC transplantation. Record the pulmonary function index including FiO2, PaO2, VT, PEEP. Participants perform the chest radiography examination before and at 24 hours, 3 Days, 7days and 1month after MSC transplantation. The severity of BPD will be further assessed by above indicators.
Short-term safety assessment of MSC transplantation by whether anaphylaxis and severe infection are observed within 24 hours after MSC transplantation. | within 24 hours after MSC transplantation
  Observed and record whether participants experience anaphylaxis including rash and anaphylactic shock within 24 hours after MSC transplantation. Also, record whether participants experience severe infection including hyperpyrexia, aggravated pulmonary inflammation and worse pulmonary function within 24 hours after MSC transplantation.
long-term safety assessment of MSC transplantation by whether intraventricular hemorrhage, periventricular leukomalacia, neurodevelopmental problems and tumor formation are observed after MSC transplantation until 24 months of corrected age. | until 24 months of corrected age
  Participants perform the cranial ultrasound to assess whether intraventricular hemorrhage and periventricular leukomalacia occur. Cranial MRI and Bayley Scale for Infant Development (BSID) are performed to assess neurodevelopment. Ultrasound and MRI examinations are performed to assess tumor formation after MSC transplantation until 24 months of corrected age.

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No